CLINICAL TRIAL: NCT06150287
Title: Effect of Probiotics on Immunosuppressive-drug-associated Diarrhea Among Renal Transplant Recipients
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: State University of New York - Upstate Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: 2044457
Record Dates: First submitted 2023-11-08; First posted 2023-11-29 (Actual); Last update posted 2024-05-13 (Actual); Status verified 2023-12

CONDITIONS: Renal Transplantation
Keywords: Probiotics; Immunosuppressive Drugs; Renal Transplantation; Diarrhea; Living Donor; Deceased Donor
MeSH Terms: conditions — Diarrhea

STUDY DESIGN:
Intervention Model Description: randomized, double-blinded, placebo-controlled, single-center pilot/exploratory trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Probiotics Group (Active Comparator): Participants will receive one probiotics capsule daily for six months immediately after the onset of post-surgical non-infectious diarrhea.
  Interventions: Other: Florajen Digestion
- Placebo Group (Placebo Comparator): Participants will receive one placebo capsule daily for six months immediately after the onset of post-surgical non-infectious diarrhea.
  Interventions: Other: Florajen Digestion

INTERVENTIONS:
Other: Florajen Digestion — Florajen Digestion is a probiotics. One probiotics capsule contains 15 billion Colony Forming Unit (CFU) of live microorganisms. No live microorganisms are present in the placebo capsules.
  Other Names: Placebo

SUMMARY:
The goal of this pilot project is to 1) examine whether oral administration of probiotics are helpful in reducing immunosuppressive drugs-associated diarrhea and adhering to the required dose of immunosuppressive drugs and 2) determine how this treatment works by examining fecal microbiome and immunological markers among living and deceased donor renal transplant recipients. The main questions it aims to answer are:

1. Does low dose probiotics effective in reducing immunosuppressive drugs-associated diarrhea?
2. Does probiotics effective in reducing inflammation?
3. Is there any connection between fecal microbiome and immunological markers?

Participants will receive one probiotics capsule or placebo capsule daily for 6 months from the onset of diarrhea post-surgically. Researchers will compare the data obtained through probiotics group and placebo group to answer the above mentioned research questions.

ELIGIBILITY:
Inclusion Criteria:

* Received living or deceased donor kidney, subjects will be monitored peri-operatively
* Presence of mild to severe diarrhea (> 3 times loose stools/day); include type 6 and 7 in the Bristol Stool Chart.
* Has been on adjusted and/or maintenance dose of calcineurin inhibitors, antimetabolites and steroid regimen. Treatment of rejection including administration of steroids, intravenous immunoglobulin/plasmapheresis, rituximab and anti- thymocytes are also acceptable in this research.

Exclusion Criteria:

* Pregnant and lactating women
* Has been receiving probiotics treatment
* Recurrence of gastrointestinal diseases including inflammatory bowel diseases, diverticulosis, irritable bowel syndrome. Had past surgical history of gastric bypass.
* Diagnosed with cancer
* Presence of infectious diarrhea, fever and high white blood cells (WBC) count. Infectious diarrhea is defined by polymerase chain reaction (PCR) negative for community acquired diarrhea panel [positive for Sapo virus, Noro virus, Clostridium difficile (positive for toxin A and B), Yersinia enterocolitica [(positive for toxin A and B) and enteropathogenic E. coli (positive Shiga toxins)].

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2024-12 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Reduction in immunosuppressive drugs-associated diarrhea | GI questionnaire and Bristol Stool Chart will be collected daily for six months from the onset of post-surgical, non-infectious diarrhea.
  Gastrointestinal (GI) questionnaire and Bristol Stool Chart will be used to measure this outcome through Chi-Square test.
Analysis of inflammatory biomarkers | Whole blood will be collected three times for six months: baseline (on the day of transplant), 3 month and six month from the onset of post-surgical, non-infectious diarrhea. three and six months
  Inflammatory biomarkers including TNF (tumor necrosis factor) superfamily proteins, IFN (interferon) family proteins, Treg cytokines and matrix metalloproteinases (MMP) [processed through Bio-Rad's Multiplex System) will be analyzed through general linear model analysis of variance (GLM ANOVA).
Association between inflammatory markers and fecal microbiome | Stool samples will be collected seven times for six months: baseline (on the day of transplant), then monthly once from the onset of post-surgical, non-infectious diarrhea.
  Fecal microbial DNA will be analyzed through 16S PCR followed by Next-Gen sequencing. Pearson correlation analysis will be performed.

CONTACTS AND LOCATIONS:
Overall Officials: Reza Saidi, Principal Investigator — State University of New York - Upstate Medical University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Roy M, Podolak T, Pankewycz O and Leftavi MR. Effect of Probiotics on Immunosuppressive Drugs Associated Diarrhea in Renal Transplant Recipients: A Practice-Based Observation. Renal Journal of Nutrition. 2018; 28:141.
- See also: Related Info — https://doi.org/10.1053/j.jrn.2018.01.012